CLINICAL TRIAL: NCT04720326
Title: Multicentre, Open-Label, Randomised, Two-Arm, Parallel-Group, Superiority Study to Assess Bioavailability and Practicability of Envarsus® Compared With Advagraf® in de Novo Liver Transplant Recipients (EnGraft)
Brief Title: Bioavailability and Practicability of Envarsus Versus Advagraf in Liver Transplant Recipients
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Edward Geissler (Other)
Collaborators: Chiesi Pharmaceuticals GmbH (Industry); Excelya (Industry)
Responsible Party: Sponsor-Investigator, Edward Geissler, Head of the Department of Experimental Surgery, University of Regensburg
Organization: University of Regensburg (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EnGraft; 2020-000796-20 (EudraCT Number)
Record Dates: First submitted 2020-12-15; First posted 2021-01-22 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Prophylaxis Against Liver Transplant Rejection
Keywords: Liver transplantation; Tacrolimus; Concentration/dose ratio; Immunosuppression
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Intervention Model Description: A dynamic allocation technique allocates participants in a 1:1 ratio to one of two treatment arms: Envarsus® tablets (test IMP) or Advagraf® capsules (comparator IMP). Pre-treatment with immediate-release tacrolimus, as well as trial site, are used as stratification factors in the treatment allocation in order to minimise sources of treatment bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Envarsus® (Experimental): Participants take prolonged-release tacrolimus tablets orally once daily and additionally receive standard-of-care immunosuppressive background therapy as per routine practice.
  Interventions: Drug: Tacrolimus Pill
- Advagraf® (Active Comparator): Participants take prolonged-release tacrolimus capsules orally once daily and additionally receive standard-of-care immunosuppressive background therapy as per routine practice.
  Interventions: Drug: Tacrolimus capsule

INTERVENTIONS:
Drug: Tacrolimus Pill — Envarsus® tablets dosed to achieve and maintain whole blood trough levels of tacrolimus within a patient-specific therapeutic range (interval of 3 ng/ml) that lies within a wider reference range of 3-12 ng/ml.
  Other Names: Envarsus
  Arms: Envarsus®
Drug: Tacrolimus capsule — Advagraf® capsules dosed to achieve and maintain whole blood trough levels of tacrolimus within a patient-specific therapeutic range (interval of 3 ng/ml) that lies within a wider reference range of 3-12 ng/ml.
  Other Names: Advagraf
  Arms: Advagraf®

SUMMARY:
Trial participants are randomised within 14 days after liver transplantation surgery in a 1:1 ratio to two alternative treatment arms containing either Envarsus® (test arm) or Advagraf® (comparator arm) as first-line calcineurin inhibitor within a standard-of-care immunosuppressive regimen. Tacrolimus blood trough levels and drug doses are monitored at regular intervals to assess drug bioavailability and the ease and accuracy of achieving the targeted blood concentration range. Dose-normalised trough level (concentration/dose ratio) is measured at 12 weeks post-randomisation as an estimate of tacrolimus bioavailability. It is hypothesised that treatment with Envarsus® will confer a superior (higher) C/D ratio after 12 weeks of therapy owing to the superior bioavailability of this galenic drug formulation (proprietary MeltDose® technology). To test whether an elevated C/D ratio is also associated with improved clinical outcomes, a range of other pharmacokinetic, efficacy and safety variables are evaluated at 10 study visits spanning a period of 3 years.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated written informed consent
2. Adult (≥18 years old) male or female
3. Recipient of a whole liver transplant from a deceased donor or a split liver transplant from a deceased or living donor
4. ABO blood type compatible with the organ donor
5. Able to swallow an oral formulation of tacrolimus in tablet or capsule form

Exclusion Criteria:

1. Multi-organ transplantation
2. Any previous organ allograft transplantation
3. Biopsy-proven acute rejection that is ongoing at the time of randomisation
4. Occurrence of post-transplant thrombosis, occlusion or stent placement in any major hepatic arteries, hepatic veins, portal vein or inferior vena cava
5. History of extra-hepatic malignancy that could not be curatively treated
6. Hepatocellular carcinoma with extra-hepatic spread or macrovascular invasion
7. Uncontrolled systemic infection
8. Requirement of life support measures such as ventilation or vasopressor agents (>20 µg/kg body weight/h) at the time of randomisation
9. Known contraindication or hypersensitivity to tacrolimus, and/or to any of the excipients listed in section 6.1 of the Summary of Product Characteristics of both Envarsus® and Advagraf®, and/or to any other macrolides
10. Ongoing, planned or foreseeable use of cyclosporine or any tacrolimus preparation other than Envarsus® or Advagraf® (except for immediate-release formulations administered before randomisation)
11. Any prolonged-release tacrolimus treatment prior to randomisation
12. Pregnant or nursing (lactating) female, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin laboratory test
13. Female of child-bearing potential, defined as physiologically capable of becoming pregnant, unless using a reliable method of contraception
14. Participation in another interventional clinical trial during the time period from randomisation to study end, if the trial is testing an Investigational Medicinal Product or if the intervention and/or follow-up requirements of the trial impede or interfere with either the objectives of EnGraft or the treatment / follow-up requirements of EnGraft
15. Any condition or factor which, in the judgement of the investigator, would place the subject at undue risk, invalidate communication with the investigator or study team, or hamper compliance with the trial protocol or follow-up schedule
16. Inability to freely give informed consent (e.g. individuals under legal guardianship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2020-12-23 (Actual); Primary Completion 2024-01-25 (Actual); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Dose-normalised blood trough level of tacrolimus (concentration/dose ratio) | 12 weeks post-randomisation
  To calculate C/D ratio, "concentration" is the blood trough level of tacrolimus measured in a blood sample collected immediately prior to drug dosing on the day of the 12-week trial visit and "dose" is the daily dose taken by the patient on the day prior to the visit. C/D ratio is measured as a surrogate for tacrolimus bioavailability (i.e. systemic exposure per mg of drug).

SECONDARY OUTCOMES:
Number of IMP dose adjustments | Until 12 weeks post-randomisation
Time to reach the first defined range in target trough level | Time period measured in days, assessed at 12 weeks post-randomisation
Number of measurements above and below the first defined range in target trough level | Time period measured in days, assessed at 12 weeks post-randomisation
Dose-normalised trough level (C/D ratio) during long-term follow-up | 1, 2 and 3 years post-randomisation
Mean tacrolimus trough level and inter-patient variability (range) of tacrolimus trough levels | 1, 2, 4 and 12 weeks post-randomisation
Inter-patient variability (range) of tacrolimus total daily dose | Until 12 weeks post-randomisation
Proportion of patients with trough levels lower, within, or higher than the standard reference range | 1, 2, 4 and 12 weeks post-randomisation
Incidence and severity of clinically-confirmed biopsy-proven acute rejection | 12 weeks and 1, 2, 3 years post-randomisation
Incidence of graft failure (defined as necessity for re-transplantation) | 12 weeks and 1, 2, 3 years post-randomisation
Incidence of death (for any reason) | 12 weeks and 1, 2, 3 years post-randomisation
Treatment failure rate (composite endpoint of biopsy-proven acute rejection, graft failure or death) | 12 weeks and 1, 2, 3 years post-randomisation
Time to treatment failure (composite endpoint of biopsy-proven acute rejection, graft failure or death) after randomisation | 3 years post-randomisation
Incidence of acute rejections requiring treatment | 12 weeks post-randomisation
Incidence of multiple rejection episodes | 12 weeks post-randomisation
Change versus baseline in laboratory measures of liver function (aspartate transaminase, alanine transaminase, alkaline phosphatase, gamma-glutamyltransferase, bilirubin, albumin, cholinesterase, INR) | 12 weeks and 1, 2, 3 years post-randomisation
Change versus baseline in laboratory measures of metabolic profile (triglycerides, HDL cholesterol, LDL cholesterol, total cholesterol, HbA1c, fasting plasma glucose) | 12 weeks and 1, 2, 3 years post-randomisation
Change versus baseline in laboratory measures of renal function (creatinine, estimated glomerular filtration rate) | 12 weeks and 1, 2, 3 years post-randomisation
Incidence and type of malignancies diagnosed in trial participants | 1, 2 and 3 years post-randomisation
Incidence and type of infections (hepatitis C virus, hepatitis B virus, cytomegalovirus, Epstein-Barr virus) experienced by trial participants | 1, 2 and 3 years post-randomisation
Degree of liver fibrosis (fibroscan or biopsy) | 12 weeks and 1, 2, 3 years post-randomisation
Incidence, type, severity, seriousness and causality of adverse events (AEs) | 3 years post-randomisation
Change versus baseline in heart rate | 3 years post-randomisation
Change versus baseline in blood pressure | 3 years post-randomisation
Change versus baseline in body weight | 3 years post-randomisation
Incidence of de novo occurrence of tremor or vision impairments | 3 years post-randomisation
Incidence of post-transplant diabetes mellitus and post-transplant hyperglycaemia | 12 weeks and 1, 2, 3 years post-randomisation
Dose-normalised trough level (C/D ratio) | 12 weeks post-transplantation
Number and doses of immunosuppressive medications (incl. other tacrolimus formulations) | At 12 weeks and after 12 weeks (if applicable)
Recurrence of primary hepatic disease | 3 years post-randomisation
Incidence of donor-specific antibodies | 12 weeks and 1, 2, 3 years post-randomisation
Continuation rate | 12 weeks post-randomisation
Incidence and time to study treatment discontinuation | 3 years post-randomisation
Incidence of patient withdrawal from the study | 3 years post-randomisation
Time to patient withdrawal from the study | 3 years post-randomisation
Reason for patient withdrawal from the study | 3 years post-randomisation

CONTACTS AND LOCATIONS:
Overall Officials: Hans J. Schlitt, MD, Principal Investigator — University Hospital Regensburg
Locations (15):
- Germany (15):
  - University Hospital Aachen, Aachen
  - Charite - University Medicine Berlin, Berlin
  - University Hospital Essen, Essen
  - University Hospital Frankfurt, Frankfurt
  - University Hospital Hamburg Eppendorf, Hamburg
  - Hannover Medical School, Hanover
  - University Hospital Heidelberg, Heidelberg
  - University Hospital Jena, Jena
  - University Hospital Schleswig-Holstein - Campus Kiel, Kiel
  - University Hospital Leipzig, Leipzig
  - University Hospital Magdeburg, Magdeburg
  - University Hospital Mainz, Mainz
  - University Hospital Muenster, Münster
  - University Hospital Regensburg, Regensburg
  - University Hospital Tuebingen, Tübingen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wohl DS, James B, Gotz M, Brennfleck F, Holub-Hayles I, Mutzbauer I, Baccar S, Brunner SM, Geissler EK, Schlitt HJ; EnGraft Trial Group. EnGraft: a multicentre, open-label, randomised, two-arm, superiority study protocol to assess bioavailability and practicability of Envarsus(R) versus Advagraf in liver transplant recipients. Trials. 2023 May 11;24(1):325. doi: 10.1186/s13063-023-07344-7. PMID 37170284